CLINICAL TRIAL: NCT04836923
Title: Home-based Physical Therapy Intervention to Decrease Frailty in Liver Transplant Candidates
Brief Title: LIFT Intervention in Liver Transplant Candidates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Daniela Ladner, Professor of Surgery - Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00213159
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Frailty; Cirrhosis; Liver Transplant
MeSH Terms: conditions — Frailty; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFT subgroup (Experimental): PT evaluation, an individualized home exercise prescription (HEP), daily text message reminders to exercise and weekly telephone check-ins with team members.
  Interventions: Behavioral: "LIver FrailTy" intervention (LIFT)
- LIFT + REAP subgroup (Experimental): PT evaluation, an individualized home exercise prescription (HEP), daily text message reminders to exercise and weekly telephone check-ins with team members. We will also employ "Realistic Effort Action Planning" (REAP), a form of personality-informed motivational interviewing in a subset of patients to potentially enhance patient engagement and adherence to the home-exercise prescription.
  Interventions: Behavioral: "LIver FrailTy" intervention (LIFT); Behavioral: "Realistic Effort Action Planning" intervention (REAP)

INTERVENTIONS:
Behavioral: "LIver FrailTy" intervention (LIFT) — Novel physical therapy intervention to decrease frailty in pre-transplant patients
Behavioral: "Realistic Effort Action Planning" intervention (REAP) — This intervention is an interactive behavioral interviewing process to engage patients in their care
  Arms: LIFT + REAP subgroup

SUMMARY:
Frailty is a significant problem in patients undergoing liver transplant and is associated with poor outcomes and survival. Hence, optimizing physical fitness and counteracting frailty is important. However, many interventions are very resource intensive and therefore not feasible.

In this study, the investigators aim to test the effectiveness of a newly designed intervention to improve frailty in liver transplant candidates. The "LIver FrailTy" intervention (LIFT) will consist of an evaluation by a physical therapist, an individualized home exercise prescription (HEP), exercise tracking using a smart phone application, daily text reminders to exercise and recurrent telephone check-ins. The investigators also aim to perform "Realistic Effort Action Planning" (REAP), which is a form of personality-informed motivational interviewing, in a subset of patients to determine if this enhances the LIFT intervention.

DETAILED DESCRIPTION:
Frailty is defined as a biologic syndrome of decreased physiologic reserve and increased vulnerability to health stressors. The concept of frailty has recently emerged as a critical determinant in the field of cirrhosis and liver transplantation. Frailty impacts pre- and post-transplant clinical outcomes, including waitlist mortality, post-transplant mortality, frequency of hospitalizations and duration of hospital admissions. Although the impact of frailty in liver transplantation has been established in the literature, there is a lack of data supporting effective interventions to decrease frailty prior to liver transplantation. Moreover, the studies that have tested interventions to improve physical function have relied on frequent supervised physical therapy sessions and access to exercise equipment that it is not financially or logistically feasible for the majority of patients. Patient engagement in PT also remains a critical barrier to overcome to decrease frailty in preparation for liver transplantation. Developing a practical and effective intervention to consistently engage patients in physical activity and decrease frailty is essential to improving clinical outcomes in the pre- and post-liver transplant setting.

The investigators goal is to pilot test a novel PT intervention to decrease frailty in pre-transplant patients. The investigators have designed a prototype "LIver FrailTy" intervention (LIFT) that includes: PT evaluation, an individualized home exercise prescription (HEP), daily text message reminders to exercise and weekly telephone check-ins with team members. The investigators will also employ "Realistic Effort Action Planning" (REAP), a form of personality-informed motivational interviewing in a subset of patients to potentially enhance patient engagement and adherence to the home-exercise prescription.

The central hypothesis is that the LIFT (+/- REAP) intervention will 1) improve adherence to recommended levels of exercise in end-stage liver disease 2) reduce pre-transplant frailty and 3) will improve pre- and post-transplant clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of liver cirrhosis being evaluated for liver transplantation in hepatology/transplant evaluation clinic
* English-speaking
* Patients with access to a smart phone (with videoconference capabilities)
* Vulnerable populations: We will include patients who are cognitively impaired due to hepatic encephalopathy and unable to consent for themselves.

Exclusion Criteria:

* Patients < 18 years of age
* Patients who require outpatient physical therapy.
* Patients without the ability to consent for themselves or through a medical power of attorney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Frailty | Every month for up to 5 years
  Frailty is described as a biologic syndrome of decreased physiologic reserve and increased vulnerability to health stressors. This outcome is measured by the Liver frailty index [LFI]. LFI is composed of 3 performance-based tests (grip strength, chair stands, and balance). There is no data to date describing the expected range of values. Higher LFI scores indicate a higher degree of frailty.
Placement on liver transplant waitlist | Every month for up to 5 years
  A clinical measure for the participant and where they are located on the liver transplant waiting list.
Clinical Outcomes - waitlist / post-transplant mortality | Every month for up to 5 years
  Measured if a patient dies while listed on the transplant waitlist or post-transplant.
Clinical Outcomes - post transplant disposition | Every month for up to 5 years
  Determined by location of patient after transplant (can be listed such as acute rehabilitation, subacute rehabilitation center, home, etc.)
Clinical Outcomes - number and duration of hospitalizations | Every month for up to 5 years
  Clinical measure for how many times a patient is hospitalized and how long those hospitalizations last.
Clinical Outcomes - liver related complications | Every month for up to 5 years
  Data collected from medical chart for liver related complications including but not limited to diagnosis of: ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome, hepatopulmonary syndrome, infection.

SECONDARY OUTCOMES:
Endurance | Every 3 months for up to 5 years
  Measured by the 4-meter walk test. Longer gait speeds suggest an increased risk of frailty.
Patient adherence | Every week for up to 5 years
  Data continuously collected via TrueCoach smart phone application to document adherence to exercise regimen. If patients are unable to appropriately track adherence on the smart phone application, this data will be collected at weekly videoconference/telephone check-ins detailed below.
Degree of hepatic encephalopathy | Every 3 months for up to 5 years
  Measured by List Sort Working Memory [LSWM] test, the Flanker Inhibitory Control and Attention [FICA], and Pattern Comparison Processing Speed Test (PCPS).
  LSWM consists of several trials wherein complementary visual and audio stimuli, presented one at a time, and participants are asked to repeat the items in order of size from smallest to largest. The raw score is the total number of lists repeated correctly. A higher score is associated with better outcomes.
  FICA examines patients' ability to inhibit visual attention to distractor arrows (flankers) and focus on a central stimulus arrow. The raw score is calculated from the response accuracy and response time over 40 trials. A higher score is associated with better outcomes.
  PCPS assesses choice reaction time by asking patients to determine whether two visual patterns are identical by "Yes" or "No". The raw score is the total correct responses out of 130. A higher score is associated with better outcomes.
Patient-reported quality of life | Every 3 months for up to 5 years
  Patient-reported quality of life is measured through a series of questionnaires a participant completes at baseline and every three months for up to five years. This outcome is measured by the National Institutes of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) Toolkit using the following validated questionnaires: Global Health Scale version 1.2, Physical Function - Short Form 8c version 2.0, Cognitive Function version 2.0, Pain Interference version 1.1, Dyspnea Severity version 1.0, Meaning and Purpose version 1.0, Fatigue version 1.0, Ability to Participate in Social Roles and Activities version 2.0. Each survey uses a 5-point Likert scale. Higher scores generally indicate poor quality of life.
Personality assessment | Every month for up to 5 years
  This outcome is measured using the Modified Midlife Development Inventory (MIDI) Personality Scale. MIDI is a list of 21 adjectives that the respondent is asked to use to rate themselves, on a four-point scale, ranging from "not at all" to "a little," "some," and "a lot."

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ladner, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thuluvath AJ, Polineni P, Morrissey S, Belfanti K, Nizamuddin M, Siddiqui O, Daud A, Simpson DC, Levitsky J, Flores AM, Duarte-Rojo A, Ladner DP. Home-based LIver FrailTy Intervention (LIFT) in Transplant Candidates: A Feasibility Study. Transplantation. 2025 Apr 1;109(4):e202-e212. doi: 10.1097/TP.0000000000005263. Epub 2024 Nov 6. PMID 40131764